CLINICAL TRIAL: NCT03678324
Title: Pre-Clinical White Matter Changes and Associated Connectivity Effects in Fabry Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: Genzyme, a Sanofi Company (Industry)
Responsible Party: Principal Investigator, Hunter Underhill, Assistant Professor of Pediatrics,, University of Utah
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Fabry MRI
Record Dates: First submitted 2018-09-06; First posted 2018-09-19 (Actual); Last update posted 2022-05-26 (Actual); Status verified 2022-05

CONDITIONS: Fabry Disease
Keywords: fabry; MRI (Magnetic resonance imaging); Fabry brain lesions
MeSH Terms: conditions — Fabry Disease | interventions — CYFIP2 protein, human

STUDY DESIGN:
Intervention Model Description: 20 patients with Fabry and 20 unaffected
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fabry (Other): Must be 18 or older and able to have an MRI.
  Interventions: Other: Functional MRI and fast bound-pool fraction imaging

INTERVENTIONS:
Other: Functional MRI and fast bound-pool fraction imaging — Use a form of MRI called fast bound-pool fraction imaging (FBFI), which is a technique better suited to capture and quantify these lesions, to study these lesions in patients with FD. In parallel, we would like to use functional MRI (fMRI) to study how these lesions alter brain function and connectivity in FD.
  Neuropsychological assessements will include Wechsler Adult Intelligence Scale, WAIS-III (Digit Span, Symbol-Digit/Coding, and Symbol Search), the Connors Continous Performance text (CPT-II). The Health Questionnaire form, the Center for Epidemiologic Studies Depression Scale (CES-D), the RAND 36-Item Health Survey.
  Other Names: fmri; FBFI; Neuropsychological assessments

SUMMARY:
The purpose of this research project is:

* to use an advanced quantitative MRI technique (FBFI) to detect and quantify brain lesion in patients with FD
* to use fMRI to identify altered brain function
* to use FBFI and fMRI together to map altered connectivity in response to brain lesions

DETAILED DESCRIPTION:
Fabry disease (FD) is a lysosomal storage disease caused by a deficiency in an enzyme that degrades components of the outer cell wall. A deficiency of this enzyme in humans has been associated with stroke. In males with FD, 6.9% have a stroke by 39 years of age. In females with FD, 4.3% have a stroke by 46 years of age.

Magnetic resonance imaging (MRI) is the main tool for studying stroke in FD. Importantly, MRI has identified other types of lesions in the brain beyond that caused by stroke. These additional lesions may herald stroke or be a different manifestation of FD in the brain. These lesions are seen in >50% of men and women with FD.

Diffusion-based imaging MRI has been the leading approach for studying these lesions in FD. However, these lesions that appear to be specific to FD are difficult to quantify, analyze, and interpret using this and other current MRI methods. The Investigators would like to use a form of MRI called fast bound-pool fraction imaging (FBFI), which is a technique better suited to capture and quantify these lesions, to study these lesions in patients with FD. In parallel, the investigators would like to use functional MRI (fMRI) to study how these lesions alter brain function and connectivity in FD. The combination of these techniques (FBFI + fMRI) will also provide us the opportunity to study brain plasticity in response to injury as Fabry disease is slowly progressive over decades allowing the brain to remodel connections to maintain function.

ELIGIBILITY:
Fabry Cohort

Inclusion Criteria:

* Have Fabry Disease
* Must be 18yrs or older

Exclusion Criteria:

* Subjects who are claustrophobic
* have metal implants
* Cannot pass the MRI safety screening questionnaire.

Unaffected Controls

Inclusion Criteria:

* Must be 18yrs or older
* unaffected with Fabry Disease
* considered healthy with no previous history of stroke, multiple sclerosis, diabetes mellitus, or other neurologic disease.

Exclusion Criteria:

* Subjects who are claustrophobic
* have metal implants
* Cannot pass the MRI safety screening questionnaire.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-01-27 (Actual); Primary Completion 2022-03-30 (Actual); Study Completion 2022-03-30 (Actual)

PRIMARY OUTCOMES:
FBFI MRI using advanced MRI technique | 6 months after enrollment closes
  advanced quantitative MRI technique (FBFI) to detect and quantify brain lesion in patients with FD
Identify difference between patients with Fabry disease and healthy controls in brain function as measured and quantified by functional MRI | 6 months after enrollment closes
  identify altered brain function
use FBFI and fMRI to map | 6 months after enrollment closes
  together to map altered connectivity in response to brain lesions

CONTACTS AND LOCATIONS:
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No
Aggregate data will be published.